CLINICAL TRIAL: NCT02753296
Title: Development and Evaluation of a Patient Fertility Preservation Decision Aid for Women With Cancer: The Cancer, Fertility and Me Research Study
Brief Title: Development and Evaluation of a Fertility Preservation Patient Decision Aid for Women With Cancer.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Sheffield (Other)
Collaborators: Yorkshire Cancer Research (Other); Weston Park Hospital Cancer Charity (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Sheffield Hallam University (Other); University of Leeds (Other); The Leeds Teaching Hospitals NHS Trust (Other); Breast Cancer Care (Charity) (Unknown); Independent Cancer Patients' Voice (Charity) (Unknown); University of Oxford (Other)
Responsible Party: Principal Investigator, Georgina Jones, Dr Georgina Jones- Reader in Social Sciences, University of Sheffield
Other Study IDs: 142491
Record Dates: First submitted 2016-04-16; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: Cancer; Fertility Preservation; Patient Decision Aid
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this research study is to develop a patient decision aid (PDA), and evaluate whether its integration within oncology services enable cancer services to effectively support and provide evidence based resources for women's fertility preservation decisions, following a diagnosis of any cancer type.

DETAILED DESCRIPTION:
Women diagnosed with cancer have to make time-pressured decisions regarding fertility preservation with specialist fertility services whilst planning their cancer treatment with oncology services. Oncologists identify a need for resources enabling them to support women's fertility preservation decisions more effectively; and women report wanting more specialist information to make these choices across service pathways. This research will develop a new evidence-based patient decision aid (PDA) to address this unmet need and evaluate its acceptability to women and services when integrated into usual cancer care pathways at the point of cancer diagnosis and treatment planning.

The objectives are to:

1. Develop a PDA for use by oncology teams to support women making fertility preservation choices, whilst having a recent cancer diagnosis.
2. Assess the validity of the PDA to support women making informed decisions about fertility preservation before starting their cancer treatment.
3. Evaluate the acceptability of the PDA to a) women making fertility preservation decisions whilst planning their cancer treatment and b) oncology and fertility health professionals supporting women's oncology and fertility treatment choices.

This research employs a series of prospective, observational surveys, employing both quantitative and qualitative methods to develop and evaluate the PDA.

Data will be collected during 5 time points:

1. Face validity stage- The purpose of this stage is to assess the face validity of the PDA from women and health professionals. Qualitative and quantitative data collection will aim to explore understanding, the purpose of the PDA, and views on its utility.
2. Evaluation Stage Baseline- Quantitative data collected from eligible women following their initial treatment planning consultation. Questionnaires are completed prior to reading the PDA.
3. Evaluation Stage Time 1- Quantitative data collected from eligible women on arrival to their appointment at the Assisted Conception Unit (ACU). For those women who decide not to attend their appointment with the fertility expert the questionnaires will be either posted or handed to them at their next oncology appointment for completion, at the same time point.
4. Evaluation Stage Time 2a- Quantitative data collected from eligible women following completion of their first round of chemotherapy.
5. Evaluation Stage Time 2b- Qualitative interview data collected from eligible women following completion of their first round of chemotherapy, and from health professionals.

ELIGIBILITY:
Inclusion Criteria: All women aged >16 of a reproductive age, with a diagnosis of any cancer, undergoing cancer treatment(s) which may impact fertility

Exclusion Criteria: Women who have started menopause/ not of a reproductive age

-

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women of a reproductive age (16yrs+), who have been diagnosed with cancer, and are undergoing or has undergone cancer treatment(s) which may impact fertility will be eligible. The sample of women will be opportunistic and identified from those women referred to the study sites.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Change in decisional conflict (Decisional Conflict Scale) | Baseline (within 3 days after initial treatment planning consultation); Time 2a- after completion of first round of chemotherapy (within 3 months after reading PDA)
  This is a 16-item measure measuring the conflict inherent in the treatment decision encountered. Scores > 37.5 on the overall scale (range 0-100) indicate high decisional conflict, which is characterised by decision delay and/or uncertainty about decision. This will be administered to women.

SECONDARY OUTCOMES:
Preparation for Decision Making Scale | Face validity stage (within one day after reading the PDA)
  This is a 10-item measure which assesses an individual's perception of how useful a DA is in preparing the respondent to communicate with their practitioner at a consultation focused on making a health decision. High scores on the overall scale (range 0-100) indicate higher perceived levels of preparation for decision making. It will be administered to women and health professionals.
Change in perception (Preparation for Decision Making Scale) | Time 1- the next oncology or fertility consultation (within one month after reading PDA)
  This is a 10-item measure which assesses an individual's perception of how useful a DA is in preparing the respondent to communicate with their practitioner at a consultation focused on making a health decision. High scores on the overall scale (range 0-100) indicate higher perceived levels of preparation for decision making. This will be administered to women.
Change in decision making readiness (The Stage of Decision Making) | Baseline (within 3 days after initial treatment planning consultation); Time 1- the next oncology or fertility consultation (within one month after reading PDA); Time 2a- after completion of first round of chemotherapy (within 3 months after reading PDA)
  This is a 6 category tool to assess the individual's readiness to engage in decision making, progress in making a choice, and receptivity to considering or re-considering options. Scores are rated 1-6 from not thinking about it at all, to considered options. This will be administered to women.
The Decisional Regret Scale | Time 2b- after completion of first round of chemotherapy (within 3 months after reading the PDA)
  This is a brief 5-item scale which measures "distress or remorse after a health care decision" using a 5-point Likert scale (1- strongly agree; 5- strongly disagree). A score of 0 on the overall scale (range 0-100) indicates no regret; scores of 100 mean high regret. This will be administered to women.
Change in health outcomes (The EQ-5D) | Baseline (within 3 days after initial treatment planning consultation); Time 2b- after completion of first round of chemotherapy (within 3 months after reading the PDA)
  This is a standardised instrument for use as a measure of health outcome. It consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. This will be administered to women.
Change in anxiety (The State Trait Anxiety Inventory) | Baseline (within 3 days after initial treatment planning consultation); Time 1- the next oncology or fertility consultation (within one month after reading PDA); Time 2a- after completion of first round of chemotherapy (within 3 months after reading PDA)
  This is a brief 6-item version used to measure of state anxiety. All items are rated on a 4-point scale (1-Almost never, 4-Almost always). Higher scores indicate greater anxiety. This will be administered to women.
Count Data | Through study completion (an average of 18 months)
  Count data will be collected of the number of DAs given to women and clinical staff, counts of use, and number of clicks on the 'Cancer, Fertility and Me' website will be recorded. In addition we will record length of oncology and fertility consultations, and length of time to fertility and cancer treatment.
Learner Verification Questionnaire | Face validity stage (within one day of reading the PDA)
  This will consist of 4 items taken from the QQ-10, which is a measure of face validity which has been used in previous studies. The 4 items will be measured on and a 5-point Likert scale (1- strongly agree; 5- strongly disagree). The questionnaire will also comprise of 3 open end questions relating to the acceptability and utility of the PDA from womens and health professionals perspective. This will be administered to women and health professionals.
Qualitative Interviews (telephone) | Face validity stage (within 1 week after reading the PDA)
  The telephone interview will take place with women and health professionals. The interview schedule will focus Learner Verification (LV) (modified from an existing LV interview schedule) to seek further clarification on answers provided on the questionnaire, and to gain more in-depth information.
Qualitative Interviews (face to face) | Time 2b- after completion of first round of chemotherapy (up to 3 months after reading the PDA)
  The interview will take place with women. The interview schedule for the face to face interviews will focus on Learner Verification (LV) (modified from an existing LV interview schedule) to explore the PDAs clarity and usefulness in planning care and making decisions between treatment options. Additional areas the interview schedule will focus on include the PDAs likelihood of use, barriers to use in practice, whether or not the women and health professionals benefit from their delivery, usefulness of the PDA in aiding service transition, and how the women used the PDA.

CONTACTS AND LOCATIONS:
Overall Officials: Georgina L Jones, D.Phil, Principal Investigator — Sheffield University
Locations (6):
- United Kingdom (6):
  - Jessop Fertility, Sheffield, South Yorkshire
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Weston Park Hospital Cancer Charity, Sheffield, South Yorkshire
  - Leeds General Infirmary, Leeds, West Yorkshire
  - Leeds Centre for Reproductive Medicine, Leeds, West Yorkshire
  - St James University Hospital, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones GL, Hughes J, Mahmoodi N, Greenfield D, Brauten-Smith G, Skull J, Gath J, Yeomanson D, Baskind E, Snowden JA, Jacques RM, Velikova G, Collins K, Stark D, Phillips R, Lane S, Bekker HL; (On behalf of the Cancer, Fertility and Me research team). Observational study of the development and evaluation of a fertility preservation patient decision aid for teenage and adult women diagnosed with cancer: the Cancer, Fertility and Me research protocol. BMJ Open. 2017 Mar 13;7(3):e013219. doi: 10.1136/bmjopen-2016-013219. PMID 28289046